CLINICAL TRIAL: NCT04882384
Title: Pericapsular Nerve Group Blocks for Hip Fractures in the Emergency Department: A Prospective, Observational, Feasibility Study
Brief Title: Pericapsular Nerve Group Block for Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobi Medical Center (Other)
Responsible Party: Principal Investigator, Anirudh Ramachandran, Co-Principal Investigator, Jacobi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-12647
Record Dates: First submitted 2021-05-08; First posted 2021-05-12 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures; Pain, Acute
MeSH Terms: conditions — Hip Fractures; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peripheral Nerve Block (PENG) (Experimental): Patients will receive the Pericapsular Nerve Group Block.
  Interventions: Procedure: Pericapsular Nerve Group Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block — This will be a peripheral nerve block.

SUMMARY:
This will be a feasibility study to see if it feasible to perform the Pericapsular Nerve Group Block for hip fractures in the Emergency Department. In addition, we will look at the efficacy of the block in these 10 patients by measuring pain scores at pre-determine time points for 16 hours.

DETAILED DESCRIPTION:
Isolated hip fractures are common and are associated with significant morbidity and mortality.1 2 The American Academy of Orthopedics provides strong evidence for peripheral nerve blocks as a safe, effective method to manage perioperative analgesia. Literature shows that peripheral nerve blocks decrease the need for opioids and its deleterious effects including respiratory depression and delirium, and can provide superior pain control when compared to parenteral analgesia.2-10 In addition to significant pain, patients with isolated hip fractures are at risk for underassessment of pain and subject to considerable delays in analgesic administration even after their pain is identified, in one study the average delay to treatment was 122 minutes.11

Ultrasound guidance has been shown to be a safe method for performing a peripheral nerve block.12 Overall, peripheral nerve blocks are a safe procedure with rare complications of nerve injury or local anesthetic toxicity.12,13

While the femoral nerve block, the "3-in-1" block, and the fascia iliaca block are popular analgesic approaches to hip fractures, they have their downsides. Literature suggests that these blocks provide inconsistent and partial analgesia.2,15, 16 A possible explanation is demonstrated by both MRI and cadaver studies that illustrate that the obturator nerve (sensory innervation) is rarely affected by these three blocks and can cause motor weakness. The potential benefit of a pericapsular nerve group (PENG) block is that its effect is sensory, while preserving motor function.

The target of the PENG block, the anterior zone of the hip, contains the highest relative concentration of sensory fibers to the hip. This part of the labrum is innervated by articular branches of the femoral nerve (FN), accessory obturator nerve (AON) and obturator nerve (ON).2 17-20 The PENG block is a novel approach described by Giron-Arango et al in 2018 as an ultrasound guided technique to target the FN, AON, and ON.2 By targeting the articular branches of these three nerves as they course between the anterior inferior iliac spine and the iliopubic eminence (IPE), the PENG block is able to provide a sensory-only blockade without causing motor weakness.2 21-23 Currently, there are case series/reports showing that the PENG block is highly efficacious for pain.

Aim/Objectives:

We intend to conduct a feasibility study among 10 emergency department (ED) patients with hip fractures to determine logistical barriers to introducing a new procedure in an ED as well as to assessing pain and efficacy of the PENG block.

Study Design:

This study will take place in the Jacobi Adult ED. This will be a 10-patient prospective, observational, feasibility study regarding the PENG block for hip fractures in adults. The emergency physician (EP) will identify 10 cognitively intact patients with hip fractures in the ED. The EP has the option to provide a standard dose of intravenous narcotics during the initial assessment if clinically warranted until radiographic confirmation of a fracture. Once a fracture has been confirmed, the research team will be contacted. The patient will be enrolled into the study if they had a pain score greater than or equal to 5/10 at triage or upon initial EP evaluation before the intravenous analgesia, if there was no pre-hospital analgesia given, and if there are no concomitant injuries. To be included into the study, the patient will be alert, oriented to person, place, and time, and must be able to demonstrate understanding of the written consent form. Patient also has to be able to indicate how much pain they are in using a visual analog pain scale, with 0 being no pain and 10 being severe pain, and be able to report any side effects experienced after administration of the nerve blockade. If the patient refuses to be in the study, it will not hinder the patient from obtaining other avenues of pain management and all other care. The pain score assessed just before the nerve block will be considered time 0. The blocks will be performed with dynamic sonographic guidance using a Sonosite X-porte machine and the curvilinear transducer using sterile technique. EP were trained on the PENG block after a workshop series consisting on a lecture and three hands- on training using a low-fidelity model. Competency was determined once the participant successfully performed the block on the low-fidelity model without intervention by the trainer. They also had to pass a three part check list, including taking consent and verbalizing aseptic technique, and scoring > 90% on a multiple choice quiz. Patients are eligible to receive standardized rescue doses of intravenous narcotics after the PENG block if they experience continued pain. Pain scores will be assessed for 16 hours at pre-determined points.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old (male or female)
* cognitive intact patients with Isolated hip fractures (both surgical and non-surgical candidates)
* displaced/non-displaced displaced/non-displaced sub-trochanteric
* displaced/non-displaced intra-trochanteric
* displaced/non-displaced femoral neck/head fractures

Exclusion Criteria:

* patient refusal
* allergy to local anesthetic
* overlying infection at injection site
* patients who cannot provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 16 hours.
  Visual Analog Pain Scale (VAS) from 0-10 with higher scores indicating worsening pain

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halperin, Principal Investigator — Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Ma YH, Wu J, Jia B, Xue JX, Wang TL. [Continuous fascia iliaca compartment block combined with oral analgesics for pre-operative pain control in elderly hip fracture patients]. Zhonghua Yi Xue Za Zhi. 2018 Mar 13;98(10):723-727. doi: 10.3760/cma.j.issn.0376-2491.2018.10.002. Chinese. PMID 29562394
- [Background] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Background] Beaudoin FL, Nagdev A, Merchant RC, Becker BM. Ultrasound-guided femoral nerve blocks in elderly patients with hip fractures. Am J Emerg Med. 2010 Jan;28(1):76-81. doi: 10.1016/j.ajem.2008.09.015. PMID 20006206
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Background] Turner AL, Stevenson MD, Cross KP. Impact of ultrasound-guided femoral nerve blocks in the pediatric emergency department. Pediatr Emerg Care. 2014 Apr;30(4):227-9. doi: 10.1097/PEC.0000000000000101. PMID 24651214
- [Background] Haines L, Dickman E, Ayvazyan S, Pearl M, Wu S, Rosenblum D, Likourezos A. Ultrasound-guided fascia iliaca compartment block for hip fractures in the emergency department. J Emerg Med. 2012 Oct;43(4):692-7. doi: 10.1016/j.jemermed.2012.01.050. Epub 2012 Apr 9. PMID 22494596
- [Background] Guay J, Parker MJ, Griffiths R, Kopp S. Peripheral nerve blocks for hip fractures. Cochrane Database Syst Rev. 2017 May 11;5(5):CD001159. doi: 10.1002/14651858.CD001159.pub2. PMID 28494088
- [Background] Hwang U, Richardson LD, Sonuyi TO, Morrison RS. The effect of emergency department crowding on the management of pain in older adults with hip fracture. J Am Geriatr Soc. 2006 Feb;54(2):270-5. doi: 10.1111/j.1532-5415.2005.00587.x. PMID 16460378
- [Background] Orebaugh SL, Kentor ML, Williams BA. Adverse outcomes associated with nerve stimulator-guided and ultrasound-guided peripheral nerve blocks by supervised trainees: update of a single-site database. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):577-82. doi: 10.1097/AAP.0b013e318263d396. PMID 22996199
- [Background] Barrington MJ, Watts SA, Gledhill SR, Thomas RD, Said SA, Snyder GL, Tay VS, Jamrozik K. Preliminary results of the Australasian Regional Anaesthesia Collaboration: a prospective audit of more than 7000 peripheral nerve and plexus blocks for neurologic and other complications. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):534-41. doi: 10.1097/aap.0b013e3181ae72e8. PMID 19916206
- [Background] Dochez E, van Geffen GJ, Bruhn J, Hoogerwerf N, van de Pas H, Scheffer G. Prehospital administered fascia iliaca compartment block by emergency medical service nurses, a feasibility study. Scand J Trauma Resusc Emerg Med. 2014 Jun 23;22:38. doi: 10.1186/1757-7241-22-38. PMID 24957807
- [Background] Swenson JD, Davis JJ, Stream JO, Crim JR, Burks RT, Greis PE. Local anesthetic injection deep to the fascia iliaca at the level of the inguinal ligament: the pattern of distribution and effects on the obturator nerve. J Clin Anesth. 2015 Dec;27(8):652-7. doi: 10.1016/j.jclinane.2015.07.001. Epub 2015 Aug 13. PMID 26277873
- [Background] Marhofer P, Nasel C, Sitzwohl C, Kapral S. Magnetic resonance imaging of the distribution of local anesthetic during the three-in-one block. Anesth Analg. 2000 Jan;90(1):119-24. doi: 10.1097/00000539-200001000-00027. PMID 10624991
- [Background] Gerhardt M, Johnson K, Atkinson R, Snow B, Shaw C, Brown A, Vangsness CT Jr. Characterisation and classification of the neural anatomy in the human hip joint. Hip Int. 2012 Jan-Feb;22(1):75-81. doi: 10.5301/HIP.2012.9042. PMID 22344482
- [Background] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Background] WERTHEIMER LG. The sensory nerves of the hip joint. J Bone Joint Surg Am. 1952 Apr;34-A(2):477-87. No abstract available. PMID 14917714
- [Background] GARDNER E. The innervation of the hip joint. Anat Rec. 1948 Jul;101(3):353-71. doi: 10.1002/ar.1091010309. No abstract available. PMID 18873153
- [Background] Gofeld M. Pericapsular nerve group (PENG) block: an ethical and academic perspective. Reg Anesth Pain Med. 2019 May 17:rapm-2019-100456. doi: 10.1136/rapm-2019-100456. Online ahead of print. No abstract available. PMID 31101728
- [Background] Acharya U, Lamsal R. Pericapsular Nerve Group Block: An Excellent Option for Analgesia for Positional Pain in Hip Fractures. Case Rep Anesthesiol. 2020 Mar 12;2020:1830136. doi: 10.1155/2020/1830136. eCollection 2020. PMID 32231802
- [Background] Kukreja P, Avila A, Northern T, Dangle J, Kolli S, Kalagara H. A Retrospective Case Series of Pericapsular Nerve Group (PENG) Block for Primary Versus Revision Total Hip Arthroplasty Analgesia. Cureus. 2020 May 19;12(5):e8200. doi: 10.7759/cureus.8200. PMID 32572357